CLINICAL TRIAL: NCT05012124
Title: Using Technology to Optimize Collaborative Care Management of Depression in Urban and Rural Cancer Centers (AKA: SUPPORTING COLLABORATIVE CARE TO OPTIMIZE PSYCHOSOCIAL ENGAGEMENT IN THE CANCER SETTING [SCOPE])
Brief Title: Using Technology to Optimize Collaborative Care Management of Depression in Urban and Rural Cancer Centers, SCOPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1121503; NCI-2021-07762 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00012892 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA244171 (NIH)
Record Dates: First submitted 2021-08-11; First posted 2021-08-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Depression; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Depression; Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic; Focus Groups; Culture Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (t-CoCM) (Experimental): Patients use the t-CoCM digital app platform and clinic care managers use the t-CoCM web-based registry platform to support delivery of collaborative care. Patient's complete surveys at baseline, 3, 6 and 9 months. Some patients also participate in an interview or focus group about their user experience with the t-CoCM digital platform. Care managers also participate in interviews regarding their experience with CoCM and the newly developed web-based platform.
  Interventions: Other: Interview or Focus Group; Other: Media/technology Intervention with collaborative care; Other: Survey Administration
- Arm II (u-CoCM) (Active Comparator): Patients receive usual care and clinic care managers deliver usual CoCM. Patients complete surveys at baseline, 3, 6 and 9 months.
  Interventions: Other: Collaborative care; Other: Survey Administration

INTERVENTIONS:
Other: Collaborative care — Receive u-CoCM
  Other Names: best practice; standard of care; standard therapy
  Arms: Arm II (u-CoCM)
Other: Interview or Focus Group — Participate in an interview or focus group
  Arms: Arm I (t-CoCM)
Other: Media/technology Intervention with collaborative care — Use t-CoCM digital platform with collaborative care
  Arms: Arm I (t-CoCM)
Other: Survey Administration — Complete surveys

SUMMARY:
This study compares the effectiveness of technology-enhanced collaborative care management (t-CoCM) to usual collaborative care management (u-CoCM) in achieving fidelity to processes of care and reducing depression symptoms in patients currently receiving cancer treatment. CoCM is a population-based, integrated care approach, where care managers, who are clinicians (typically clinical social workers), deliver behavioral treatments, coordinate psychosocial care, monitor outcomes, and adjust treatment with the input of a psychiatric consultant. The use of t-CoCM may improve the treatment of depression and improve patient outcomes and quality of life.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (t-CoCM): Patients use the t-CoCM digital app platform and clinic care managers use the t-CoCM web-based patient registry platform to support delivery of collaborative care. Patients complete surveys at baseline, 3, 6 and 9 months. Some patients also participate in an interview or focus group about their user experience with the t-CoCM digital platform. Care managers also participate in interviews or focus groups regarding their experience with CoCM and the newly developed web-based platform.

ARM II (u-CoCM): Patients receive usual care and clinic care managers deliver usual CoCM. Patients complete surveys at baseline, 3, 6 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving active treatment (surgery, chemotherapy, immunotherapy, targeted therapy, stem cell transplant, hormone therapy, radiation therapy) for a malignancy
* >= 18 years old
* Participants must be ambulatory for clinical care visits
* Clinically significant depression (Patient Health Questionnaire-9 (PHQ-9) >= 10 with at least one cardinal symptom > 1)
* Access to smartphone, tablet, or computer with internet access; or landline

  * Patients who do not have a smartphone will be offered assistance in obtaining a free smartphone through the government-sponsored Lifeline Phone Program for low-resourced individuals

Exclusion Criteria:

* Advanced cancer or other condition that limits remaining life expectancy to less than 9 months
* Already engaged in or needing immediate specialty mental health care e.g., for bipolar disorder or schizophrenia
* Inability to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Level of treatment engagement (collaboration & coordination of care) | Baseline to 12 months
  Follow-up contacts (in person, phone or video) documented in patient registry and electronic health record (EHR). Case reviews with consulting study psychiatrist. Total time spent interacting with patients documented by the care manager in the patient registry.
Use of depression patient-reported outcomes for measurement-based care | Baseline to 12 months
  Patient-reported depression measure (PHQ-9) score collected (in person or remotely) and entered into patient registry.
Adherence to guideline-level depression treatment | Baseline to 12 months
  Antidepressant treatment: Achieving therapeutic dose for at least 6 weeks. Dosage and adherence recorded in the patient registry and EHR, and self-reported medication data requested at 3, 6, and 9 month outcome assessments.
Change in depression severity | Baseline, 3, 6, and 9 months
  The Symptom Checklist (SCL)-20 depression scale contains the 20 items from the SCL-90 that relate specifically to depressive symptoms.

SECONDARY OUTCOMES:
Change in patient-centered shared decision-making score | 3, 6, and 9 months
  The 9-item Shared Decision-Making Questionnaire (SDM-Q-9) will be adapted and administered.
Change in anxiety severity | Baseline, 3, 6, and 9 months
  The SCL-10 contains the 10 items from the SCL-90 that relate specifically to anxiety symptoms.
Change in patient-reported depression severity | Baseline to 12 months
  Self-report Patient Health Questionnaire (PHQ-9) collected from patient registry and patient medical records.
Change in patient-reported anxiety severity | Baseline to 12 months
  Self-report Generalized Anxiety Disorder questionnaire (GAD-7) collected from patient registry and patient medical records.
Change in health-related quality of life global scales and subscales | Baseline, 3, 6, and 9 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 - Functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures.
Change in functional status | Baseline, 3, 6, and 9 months
  The Sheehan Disability Scale (SDS) was developed to assess functional impairment in three inter-related domains; work/school, social, and family life.
Change in patient impression of change and satisfaction with care | 3, 6, and 9 months
  The Patient's Global Impression of Change (PGIC) and satisfaction with care (7- point Likert) scales.
Change in health services utilization | Baseline, 3, 6, and 9 months
  Cornell Services Index (CSI), measures the quantity and characteristics of health services used in the past 3 months.
Change in environmental reward score | Baseline and 6 months
  Environmental Reward Observation Scale (EROS) measures self-rated environmental reward and response-contingent positive reinforcement.
Change in Instrumental Support: patient's perception of available support | Baseline and 6 months
  NIH Toolbox Instrumental Support Survey measures patient's perceived availability of people who can provide functional aid to help them complete daily tasks.
Change in Alcohol, Smoking, and Substance Use | Baseline and 6 months
  Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) documents psychoactive substance use and related problems in patients.
Change in Daily Alcohol Use | Baseline and 6 months
  Daily Drinking Questionnaire (DDQ) measures the quantity and frequency of participant's alcohol use.
Change in Cannabis Use | Baseline, 3, 6, and 9 months
  Self-report survey about patient's reasons, routes of administration, and frequency of cannabis use.
Change in Use of Complementary and Alternative Therapy Use | Baseline and 6 months
  Self-report survey about patient's recent use of complementary and alternative therapies.
Patient's experience using the new technology | Survey: 6 Months; Interview/focus group: between 6-12 months
  Self reported survey; and for a subset of participants, an interview or focus group
Care Managers experience using the new technology | Up to 5 years
  Interview or focus group of care managers
Care manager (CM) satisfaction with Collaborative Care Management (CoCM) of depression | At the end of the study or when a Care Manager leaves their role (Up to 5 years)
  Measures CM satisfaction with implementation of CoCM.
Oncology provider's perception of patient's adherence to cancer treatment | After the patient is sent their 9 Month survey. Oncologists may participate on behalf of multiple patients for a period of up to 3 years)
  The patient's primary oncology provider will complete a standardized questionnaire to report delays or disruptions encountered in their planned cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse R. Fann, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - MultiCare Regional Cancer Center - Gig Harbor, Gig Harbor, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT05012124/ICF_000.pdf